CLINICAL TRIAL: NCT05540886
Title: CLEAN FRONTLINE CAMBODIA A Stepped Wedge Cluster Trial of an Environmental Hygiene Educational Intervention Across Thirteen Cambodian Hospitals
Brief Title: CLEAN Frontline: A Stepped Wedge Cluster Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: National Institute of Public Health, Cambodia (Other Government); WaterAid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: 26637
Record Dates: First submitted 2022-09-01; First posted 2022-09-15 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2022-02

CONDITIONS: Hospital Infections; Environment, Controlled; Infection Control
MeSH Terms: conditions — Cross Infection

STUDY DESIGN:
Intervention Model Description: This is a randomised cluster controlled trial using a stepped-wedge random allocation. At four distinct time points, 13 hospitals will receive the educational intervention. The unit of analysis is high frequency touches sites in the three wards of interest in each of the study hospitals.
Who Masked: Outcomes Assessor
Masking Description: Staff who clean will not be blinded as this is not possible. An independent team (not involved in the delivery of the training) will collect monthly primary outcome data from pre-agreed hospital sites. The laboratory team processing the primary outcomes are also blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Standard practices are expected at hospitals before the education intervention is deployed
- Intervention (Experimental): The main intervention - the training of trainers/champions (ToT) will be delivered to selected facility "cleaning champions" from three or four hospitals within a certain month. Four sets of ToT are expected to happen during the study period.
  Interventions: Behavioral: TEACH CLEAN

INTERVENTIONS:
Behavioral: TEACH CLEAN — The intervention is primary a training facility cleaning champions to educate and supervise other existing facility cleaners with environmental hygiene responsibilities - training of trainers (ToT).
  The training content includes as much as possible the seven contextualized modules of TEACH CLEAN training package (CLEAN BOX): i) Introduction to Infection Prevention and Control, ii) Personal hygiene and dress code, iii) Hand hygiene, iv) Personal protective equipment, v) Housekeeping/control of environment, vi) Waste handling, and vii) Linen handling.
  Facility training will occur in three selected wards: i) maternity ward, including labour and post-natal rooms, ii) medicine ward, iii) and medicine ward.
  There is also supervision stage that refers to ongoing mentorship of cleaning champions by the local partner while they educate and supervise existing facility cleaners with environmental hygiene responsibilities.
  Arms: Intervention

SUMMARY:
Environmental hygiene is a key component of infection prevention in healthcare, and a driver of healthcare associated infections. Staff who clean in many low resource countries receive no formal training on cleaning, waste disposal and linen handling. This issue has been execrated by the COVID-19 pandemic. The only recommended training on environmental hygiene for low resourced facilities, TEACH CLEAN, uses a training of trainers model. A selected cadre "champions" which in turn train their peers with responsibilities on environmental hygiene at the facility level. Early pilot data to test its effectiveness of this training package are very promising.

The main objective is to evaluate the effectiveness of an environmental cleaning bundle to improve microbiological cleanliness in Cambodian hospitals.

The latest TEACH CLEAN will be implemented across all hospitals (13) of three provinces in Cambodia. A stepped wedge randomised trial will be used to evaluate the effectiveness of TEACH CLEAN to improve microbiological cleanliness in Cambodian hospitals. All facilities will receive the intervention. Hospitals are arranged in groups of three or four based on the randomisation with staggered commencement dates of the intervention at four distinct time points. The design will include ten months of data collection. We expect one month gap between the training of champions and the training of staff at the facility level. The main outcome is microbiological cleanliness (<2.5 cfu/cm2 = clean ; ≥2.5 cfu/cm2 = not clean) measured using a non-specific agar on one side for measuring total Aerobic Colony Counts (ACC/cm2). With 30 sampling sites in each hospital and with a pre-training cleanliness proportion ranging from 30% to 50% will give us over 85% power to detect a 10% absolute post-intervention increase in cleanliness.

Evidence from this trial will contribute to future policy and practice guidelines about hospital environmental hygiene and ultimately reduce healthcare associated infections. This would be the first randomised trial on environmental hygiene in low resource settings.

ELIGIBILITY:
Inclusion criteria for surfaces sites selected for primary outcome measurement

* Surfaces within the patient zone which frequently touched surfaces of the targeted wards: maternity, pediatric and general medicine

Exclusion Criteria:

* Surfaces outside the patient zone
* Surfaces not in the wards of interest

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 390 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Microbiological cleanliness | Data is collected monthly during the study period from each of the study sites. Because this is a stepped wedge trial with four steps, the data collection period referring to the pre-training/intervention period varies between 2 and 7 months. Whereas the
  The unit of measurement is high touch surfaces within the patient zone in each ward. Proportion of microbiological cleanliness (<2.5 cfu/cm2 = clean ; ≥2.5 cfu/cm2 = not clean) will be calculated for each cluster as the number of sites with <2.5 cfu/cm2 out of the 30 sites sampled per period/month.

OTHER OUTCOMES:
Changes over time in microbiological cleanliness | Data is collected monthly during the study period from each of the study sites. Because this is a stepped wedge trial with four steps, the data collection period referring to the pre-training/intervention period varies between 2 and 7 months. Whereas the
  The unit of measurement is high touch surfaces within the patient zone in each ward. Proportion of microbiological cleanliness (<2.5 cfu/cm2 = clean ; ≥2.5 cfu/cm2 = not clean) will be calculated for each cluster as the number of sites with <2.5 cfu/cm2 out of the 30 sites sampled per period/month.

CONTACTS AND LOCATIONS:
Locations (1):
- National Insitute of Public Health, Phnom Penh, Cambodia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gon G, Ma S, Aiken AM, Dancer SJ, Graham WJ, Nash S, Nov V, Mao S, Sarpong B, Pepper M, Vong S, Tang V, Thompson J, Por I. Impact of a multicomponent training intervention (Clean FrontLine) on microbiological cleanliness in Cambodian referral hospitals: a multicentre, stepped-wedge, cluster-randomised trial. Lancet Microbe. 2025 Dec 10:101262. doi: 10.1016/j.lanmic.2025.101262. Online ahead of print. PMID 41389803

DOCUMENTS (2):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form: Study Protocol (2022-02-07): https://cdn.clinicaltrials.gov/large-docs/86/NCT05540886/Prot_SAP_ICF_001.pdf
  • Statistical Analysis Plan: Analysis Plan (2023-06-06): https://cdn.clinicaltrials.gov/large-docs/86/NCT05540886/SAP_002.pdf